CLINICAL TRIAL: NCT06779383
Title: Effect of Pilates Mat Exercises Training on Functional Performance in Middle Age Obese Women: Randomized Controlled Trial
Brief Title: Pilates Mat Exercises Training on Functional Performance in Middle Age Obese Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Abdelkhalek, assistance professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pilates exercise on obesity
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: sixty obese women patients (ages 45-55 years old) with a body mass index (BMI) 30 -34.9 kg/m2.Women will be randomly assigned into experimental group(Pilates) or control group, (3 times/week, 60 min/session) their age from 45 to 55 yrs. The Pilates exercises were performed on mats. The functional performance on one-leg stance (OLS), five-times-sit-to-stand (STS) and 6-min walk (6 MW) tests was evaluated before and after the 12-week Pilates training or control follow-up period.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates mat exercises (Experimental): 30 obese women patients Pilates exercises were performed on mats. The functional performance on one-leg stance (OLS), five-times-sit-to-stand (STS) and 6-min walk (6 MW) tests was evaluated before and after the 12-week Pilates training
  Interventions: Other: pilates mat exercises
- control (No Intervention): 30 obese women patients (ages 45-55 years old) with a body mass index (BMI) 30 -34.9 kg/m2.Women will be randomly assigned into control group

INTERVENTIONS:
Other: pilates mat exercises — The Pilates exercises were performed on mats. The functional performance on one-leg stance (OLS), five-times-sit-to-stand (STS) and 6-min walk (6 MW) tests was evaluated before and after the 12-week Pilates training or control follow-up period.
  Arms: pilates mat exercises

SUMMARY:
• Aim of the study: This study will aim to investigate the effects of a 12-week Pilates-mat exercise program on the functional performance in middle age obese women.

Materials and Methods:

sixty obese women patients (ages 45-55 years old) with a body mass index (BMI) 30 -34.9 kg/m2.Women will be randomly assigned into experimental group(Pilates) or control group, (3 times/week, 60 min/session) their age from 45 to 55 yrs. The Pilates exercises were performed on mats. The functional performance on one-leg stance (OLS), five-times-sit-to-stand (STS) and 6-min walk (6 MW) tests was evaluated before and after the 12-week Pilates training or control follow-up period.

DETAILED DESCRIPTION:
One of the major public health challenges of the 21st century is obesity. In simple terms, obesity is an excessive increase in fat mass. Since the 1980s, its prevalence has tripled in many countries and the population with weight excess continues to grow at an alarming rate. Obesity impacts on morbidity, disability, activities of daily living and increases the risk of developing cardiovascular disease. (Ghiotto et.al 2022). In addition, Obesity is associated with a risk of decrease in functional capacity and muscle strength. (Lakhdar et. al 2023).

Pilates exercises consist of stretching and endurance movements performed within the range of joint motions at a regulated pace with concentration and deep breathing. This workout is a novel approach to physical training that involves a combination of strength, stretching, and respiratory and muscular motions. It aims to build muscle, enhance cardiac and respiratory indices, and promote weight loss. In contrast to conventional resistance exercises, in which individual muscle groups are trained, Pilates exercises require the activation and coordination of several muscle groups. (Hushmandi et .al 2023).

ELIGIBILITY:
Inclusion Criteria:

* women

  * BMI between 30 to 34.9 kg/m2
  * Age will range from 45-55 years old.

    1. Exclusion criteria

Exclusion Criteria:

* Cardiac diseases

  * Liver diseases
  * Hypertension
  * Musculoskeletal disease

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
  * BMI between 30 to 34.9 kg/m2
  * Age will range from 45-55 years old.
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
BMI | at baseline and after three month
  body mass index
OLS | at baseline and after three month
  One-leg stance
STS | at baseline and after three month
  Five-times-sit-to-stand
6 MW | at baseline and after three month
  6-min walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Abdelkhalek, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No